CLINICAL TRIAL: NCT00176163
Title: Supporting Effect of Dronabinol on Behavioral Therapy in Fibromyalgia and Chronic Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Central Institute of Mental Health, Mannheim (Other); University of Mannheim (Other); Academic City Hospital, Germany (Other); BG Trauma Center Ludwigshafen (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: kfg107
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2005-09

CONDITIONS: Fibromyalgia; Back Pain
Keywords: Fibromyalgia; Back pain; Behavior Therapy; Operant learning; Tetrahydrocannabinol
MeSH Terms: conditions — Fibromyalgia; Back Pain | interventions — Dronabinol

INTERVENTIONS:
Behavioral: Operant behavioral treatment; Drug: THC

SUMMARY:
It is known, that a so called "pain memory" usually evolves in chronic pain syndromes which both aggravates the disorder and modifies the patients pain perception. Thus, the principal object of pain therapy is to "delete" this dysfunctional pain memory. The combination of medication, physiotherapy and psychological therapy seems to be the most effective treatment. This study investigates the effect of a concomitant Dronabinol medication (Cannabinoid) on the effectiveness of behavioral therapy. It is hypothesized that the combination of behavioral therapy and Dronabinol will be most effective in deleting the pain memory.

DETAILED DESCRIPTION:
This study investigates the combination of operant behavioral treatment and Cannabinoid medication in patients with fibromyalgia and patients with back pain. It is well known that cannabinoids (THC) accelerate learning processes. It is assumed that the combination of both treatments may exert an synergetic effect. A low dose of THC is used, which ist not expected to have direct analgetic effects. The study also investigates genetic determinants of both disorders and the response to treatment, respectively.

The patients will be randomly assigned to one of four groups: Behavioral therapy and Dronabinol, behavioral therapy and placebo, behavioral therapy only, standard medical therapy. Patients will attend 12 weekly group-sessions (6-8 patients) of behavioral therapy. Behavioral therapy sessions will include training in reducing pain behaviour and establishing active and "healthy" behaviour instead. There will be weekly medical safety visits, in which the patients receive medication and undergo a physical examination (blood and urine samples).

Patients will be evaluated before and after behavioral therapy and will be followed for an additional 6- and 12-months phase. The outcome variables will be recorded by the use of interviews and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Fibromyalgia meeting ACR-criteria
* Diagnosis of chronic back pain
* Pain duration exceeding 3 months
* Age between 18 and 70 years
* The patient has been informed about the study, understood the information and signed the informed consent form

Exclusion Criteria:

* Tumors, fractures and heavy osteoporosis
* Secondary back pain at arthrosis or degenerative scoliosis
* Radicular back pain
* Other pain syndrome is main problem
* Opiate medication > 60mg morphine per diem
* Addiction (drugs, alcohol, medicaments)
* Cardiac insufficiency > NYHA II
* Exercise induced dyspnea, Angina pectoris A detailed version of exclusion criteria: see study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2005-08; Study Completion 2009-05

PRIMARY OUTCOMES:
Impairment by pain

SECONDARY OUTCOMES:
Pain intensity
physical function and emotional state assessed by questionnaires
number of serious adverse events
subjective rating of improvement by therapy
subjective rating of therapy effectiveness
therapy satisfaction rated by patient

CONTACTS AND LOCATIONS:
Overall Officials: Justus Benrath, MD, PhD, Principal Investigator — Heidelberg University

REFERENCES:
- [Derived] Finnern MM, Kleinbohl D, Flor H, Benrath J, Holzl R. Deconstructing chronicity of musculoskeletal pain: intensity-duration relations, minimal dimensions and clusters of chronicity. Scand J Pain. 2018 Jul 26;18(3):363-377. doi: 10.1515/sjpain-2018-0021. PMID 29870396